CLINICAL TRIAL: NCT06465979
Title: Perception of Speech in Context by Listeners With Healthy and Impaired Hearing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Christian Stilp, Associate Professor, Marquette University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4824; R01DC020303 (NIH)
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hearing; Hearing Loss
Keywords: speech perception; hearing
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech perception experiments (Experimental): This arm involves experiments wherein participants listen to speech played at comfortable volumes and respond by indicating what they heard either in open-ended form or by choosing among a set of options displayed on a computer.
  Interventions: Behavioral: Speech Manipulation

INTERVENTIONS:
Behavioral: Speech Manipulation — The acoustic properties of speech sounds will be modified in two main ways. The first way is to introduce gradual changes to the perceived articulation of the target speech sound, such as changing from "sh" to "s" by various types of signal processing and filtering. The second type of change is to modify acoustic properties of the sounds that immediately precede the target speech sound, such as changing the speaking rate or its frequencies composition.

SUMMARY:
Recognition of speech sounds is accomplished through the use of adjacent sounds in time, in what is termed acoustic context. The frequency and temporal properties of these contextual sounds play a large role in recognition of human speech. Historically, most research on both speech perception and sound perception in general examine sounds out-of-context, or presented individually. Further, these studies have been conducted independently of each other with little connection across labs, across sounds, etc. These approaches slow the progress in understanding how listeners with hearing difficulties use context to recognize speech and how their hearing aids and/or cochlear implants might be modified to improve their perception. This research has three main goals. First, the investigators predict that performance in speech sound recognition experiments will be related when testing the same speech frequencies or the same moments in time, but that performance will not be related in further comparisons across speech frequencies or at different moments in time. Second, the investigators predict that adding background noise will make this contextual speech perception more difficult, and that these difficulties will be more severe for listeners with hearing loss. Third, the investigators predict that cochlear implant users will also use surrounding sounds in their speech recognition, but with key differences than healthy-hearing listeners owing to the sound processing done by their implants. In tandem with these goals, the investigators will use computer models to simulate how neurons respond to speech sounds individually and when surrounded by other sounds.

DETAILED DESCRIPTION:
Participants in this study listen to speech played at a comfortable volume and respond by indicating what they heard, either in open-ended form or by choosing among a set of options displayed on a computer. They are seated inside a sound booth and complete the task at their own pace, with little intervention needed from the experimenter. Upon arrival at the lab, participants are given a brief description of the topic of the research (how earlier sounds influence our perception of later speech sounds) and are presented with a detailed informed consent form. Their demographic information is collected and then the experiment is demonstrated. Breaks are offered between testing blocks, which last about 10-15 minutes each.

The main differences in the protocol consist of the various stimulus manipulations, which are designed to specifically control aspect of the voice that the participant hears. For example, the sound can be manipulated to emphasize higher or lower frequencies, or be spoken relatively slowly or quickly, or manipulated to sound degraded, as if the participant has a hearing loss. In all occasions, the manipulations are signaled to the participant. The outcome measure typically consists of the pattern of word identification, and specifically how that pattern changes depending on acoustic properties of the sounds heard before the target word.

Additional comparison measurements are taken of the participant's ability to hear and repeat words or sentences in background noise.

Once an experiment is ready to launch, participants are randomly assigned to different testing conditions ("interventions"). But in most of the planned experiments, participants complete identical protocols, except that the specific ordering of many speech stimuli is randomized within the testing session. After the participant completes all of the testing blocks, they are debriefed about the full nature of the study, the hypotheses and the larger scope of the project in the context of speech communication.

ELIGIBILITY:
Inclusion Criteria:

* Be able to recognize spoken words in English
* Be a competent speaker of north American English
* Be an adult between the age of 18 to 65 years
* Have normal audiometric thresholds below 25 decibels hearing loss (dB HL) at frequencies between 250 and 8000 Hz OR have audiometric thresholds not exceeding 40 dB HL at frequencies between 250 and 8000 Hz OR have audiometric thresholds not exceeding 55 dB HL at frequencies between 250 and 8000 Hz OR use a cochlear implant
* Lack language-learning or other cognitive disabilities

Exclusion Criteria:

* Inability to recognize spoken words in English
* Not a competent speaker of north American English
* Be younger than 18 years of age
* Be older than 65 years of age
* Have normal audiometric thresholds exceeding 25 dB HL at frequencies between 250 and 8000 Hz OR have audiometric thresholds exceeding 40 dB HL at frequencies between 250 and 8000 Hz OR have audiometric thresholds exceeding 55 dB HL at frequencies between 250 and 8000 Hz
* Language-learning or other cognitive disabilities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Speech categorization | "Post-treatment" where "treatment" is the systematic manipulation of speech sounds. Speech categorization will be evaluated during the main part of the testing. Outcomes will be assessed and data reported through study completion, an average of 1 year
  The participant sits inside a double-walled sound booth. They are seated at a table that contains a computer monitor and a mouse. A single utterance is played over headphones or through a loudspeaker directly in front, and the participant indicates what they thought the utterance was by selecting among various options on the screen using the mouse. During a single block of trials there are between 60 and 160 sounds, depending on the exact experiment. Ordering of stimuli within the block is randomized. That testing block may be repeated multiple times so that the proportion of responses for each sound-response pair can be estimated reliably and precisely. Completion and advancement of trials is at the participant's own pace. Each testing block takes between 4 and 15 minutes.

SECONDARY OUTCOMES:
Speech recognition | "Post-treatment" where "treatment" is the systematic manipulation of speech sounds. Word recognition will be evaluated during the main part of the testing. Outcomes will be assessed and data reported through study completion, an average of 1 year
  The participant sits inside a double-walled sound booth. They are seated at a table that contains a computer monitor and a mouse. Recorded sentences are played over headphones or through a loudspeaker directly in front, and the participant indicates what they thought the utterance was by typing their response or repeating the sentence aloud. During a single block of trials there are 50 words. Ordering of words within the block is randomized. Completion and advancement of trials is at the participant's own pace. Each testing block takes between 6 and 15 minutes.
Audiometric threshold testing | Baseline
  The participant sits inside a double-walled sound booth. Under headphones, they listen for soft tones played by an audiometer. The experimenter controls the timing, frequency and intensity of those tones to find the lowest sound intensity where the participant can detect the tone. Thresholds for sound detection are recorded for octave frequencies between 250 Hz and 8000 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Stilp, PhD, Principal Investigator — Marquette University
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Marquette University, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made public for purposes of resource sharing and demonstration of research method / analysis. These data, materials used to generate stimuli, and materials used to perform statistical analysis will be made freely available on the Open Science Framework website.
Supporting Information: SAP
Time Frame: Data will be made available to all upon acceptance of manuscripts for publication in scholarly journals. Data will be available for a period of at least 10 years or the retirement of both investigators, which is not anticipated to be less than 15 years.
Access Criteria: Materials will be made public to all upon acceptance of manuscripts for publication in scholarly journals.